CLINICAL TRIAL: NCT03650049
Title: Food Protein-induced Enterocolitis Syndrome (FPIES) in 14 Children
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: R2016-20
Record Dates: First submitted 2018-08-22; First posted 2018-08-28 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Allergy; Pediatric Disorder
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Food protein-induced enterocolitis syndrome (FPIEES) is a particular non-Immunoglobulin E-mediated food allergy.

A retrospective descriptive single-center study was conducted. Subjects included were children with acute FPIES who consulted the allergy department of the Nancy Regional University Hospital between November 2013 and June 2016.

DETAILED DESCRIPTION:
As it is a descriptive study, the Primary Outcome is not a Measure. Therefore it is not possible to include the name of the measurement or measurement tool used to assess the measure in the primary outcome measure title.

ELIGIBILITY:
Inclusion Criteria:

* Child from 0 to 17 years with acute FPIES

Exclusion Criteria:

-

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with acute FPIES who consulted the allergy oupatient clinic of the Nancy Regional University Hospital between November 2013 and June 2016.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
symptoms due to FPIES | from november 2013 to june 2016
  description of symptoms due to acute FPIES and chronic FPIES